CLINICAL TRIAL: NCT02456051
Title: Role of Adrenomedullin in Early Diagnosis of Pancreatic Cancer in New Onset Diabetes Patients
Brief Title: Pancreatic Cancer Can be Detected by Adrenomedullin in New Onset Diabetes Patients
Acronym: PaCANOD
Status: Terminated | Type: Observational
Why Stopped: enrollment was terminated because of the poor recruitment rate
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Laura Antolino, MD, University of Roma La Sapienza
Other Study IDs: 3463_2014_D'Angelo
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Adult-Onset; Diabetes Complications; Carcinoma, Pancreatic Ductal; Pancreatic Neoplasm
Keywords: Pancreatic Carcinoma; New-Onset Diabetes; Adrenomedullin; Early Diagnosis; Biological Markers
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Complications; Carcinoma, Pancreatic Ductal; Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- High AM: Newly diagnosed diabetic patients with high Adrenomedullin serum levels
- Low AM: Newly diagnosed diabetic patients with low Adrenomedullin serum levels

SUMMARY:
Pancreatic Cancer is a leading cause of cancer-related death. To date, only one fifth of patients at diagnosis is presented resectable because the diagnosis is often delayed making the 5-year survival of this disease globally less than 5%. An early diagnosis in these patients is currently not possible given the economic disadvantages of a population-wide screening. New evidences identify patients with new-onset diabetes as a subgroup of patients at high risk of developing this disease (RR 5:38). In a subset of these patients a mediator secreted by the tumor, the Adrenomedullin, could be responsible for the onset of diabetes. Our goal is therefore to assess the different impact of Pancreatic Cancer depending on Adrenomedullin values in patients with newly diagnosed diabetes mellitus.

DETAILED DESCRIPTION:
The study is defined as prospective observational. The research project involves the recruitment prospectively for all consecutive patients aged between 45 and 75 years receiving a new diagnosis of diabetes, according to the criteria established by the American Diabetes Association (ADA) (fasting glucose greater than or equal 126 mg / dl, or random blood glucose greater than or equal to 200 mg / dl, or glycated hemoglobin greater than or equal to 6.25%). The recruitment will take place at the Sant'Andrea Hospital. The suitability of a subject to be included in the study will be evaluated by medical history, physical examination and any further investigations carried out by a medical researcher of the team, according to the inclusion and exclusion criteria. The research team will be multidisciplinary, translational, composed of medical specialists belonging to the departments of General Surgery, Internal Medicine, Diabetology and Occupational Medicine. An informed consent will be mandatory for the recruitment in the study. At recruitment Adrenomedullin serum levels will be recorded along with every relevant clinical and laboratory data. An annual telephone follow-up will be applied and if necessary the patient will benefit of an outpatient examination. A sample size of 440 patients will achieve 80% power to detect a statistically significant difference. The 3 years clinical follow-up will allow the detection of symptoms and signs that could be related to the presence of a pancreatic mass (jaundice, pain, weight loss), further investigations will follow in such cases to confirm Pancreatic cancer diagnosis and proceed to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 75 years
* Diagnosis of diabetes mellitus made within the two years preceding the date of observation (new onset diabetes)
* Adherence to the study documented the voluntary signing of an informed consent
* Availability to follow a telephone follow-up

Exclusion Criteria:

* Remote medical history (> 2 years) positive for diabetes mellitus
* Previous history of malignancy
* Pregnancy
* Renal Failure
* Documented diabetic microangiopathy
* Sepsis

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients newly diagnosed of diabetes, according to the criteria established by the American Diabetes Association (ADA) (fasting glucose greater than or equal to 126 mg/dl, or random blood glucose greater than or equal to 200 mg/dl, or glycated hemoglobin greater than or equal to 6.5%)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Pancreatic cancer diagnosis | 3 years

SECONDARY OUTCOMES:
Mortality | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Antolino, MD, Principal Investigator — Università Sapienza di Roma
Locations (1):
- Università Sapienza di Roma, Azienda Ospedaliera Sant'Andrea, Roma, Italy

REFERENCES:
- [Background] Poruk KE, Firpo MA, Adler DG, Mulvihill SJ. Screening for pancreatic cancer: why, how, and who? Ann Surg. 2013 Jan;257(1):17-26. doi: 10.1097/SLA.0b013e31825ffbfb. PMID 22895395
- [Background] Chari ST, Leibson CL, Rabe KG, Timmons LJ, Ransom J, de Andrade M, Petersen GM. Pancreatic cancer-associated diabetes mellitus: prevalence and temporal association with diagnosis of cancer. Gastroenterology. 2008 Jan;134(1):95-101. doi: 10.1053/j.gastro.2007.10.040. Epub 2007 Oct 26. PMID 18061176
- [Background] Yachida S, Jones S, Bozic I, Antal T, Leary R, Fu B, Kamiyama M, Hruban RH, Eshleman JR, Nowak MA, Velculescu VE, Kinzler KW, Vogelstein B, Iacobuzio-Donahue CA. Distant metastasis occurs late during the genetic evolution of pancreatic cancer. Nature. 2010 Oct 28;467(7319):1114-7. doi: 10.1038/nature09515. PMID 20981102
- [Background] Huxley R, Ansary-Moghaddam A, Berrington de Gonzalez A, Barzi F, Woodward M. Type-II diabetes and pancreatic cancer: a meta-analysis of 36 studies. Br J Cancer. 2005 Jun 6;92(11):2076-83. doi: 10.1038/sj.bjc.6602619. PMID 15886696
- [Background] Ben Q, Xu M, Ning X, Liu J, Hong S, Huang W, Zhang H, Li Z. Diabetes mellitus and risk of pancreatic cancer: A meta-analysis of cohort studies. Eur J Cancer. 2011 Sep;47(13):1928-37. doi: 10.1016/j.ejca.2011.03.003. Epub 2011 Mar 31. PMID 21458985
- [Background] Chari ST, Leibson CL, Rabe KG, Ransom J, de Andrade M, Petersen GM. Probability of pancreatic cancer following diabetes: a population-based study. Gastroenterology. 2005 Aug;129(2):504-11. doi: 10.1016/j.gastro.2005.05.007. PMID 16083707
- [Background] Pannala R, Leirness JB, Bamlet WR, Basu A, Petersen GM, Chari ST. Prevalence and clinical profile of pancreatic cancer-associated diabetes mellitus. Gastroenterology. 2008 Apr;134(4):981-7. doi: 10.1053/j.gastro.2008.01.039. Epub 2008 Jan 18. PMID 18395079
- [Background] Aggarwal G, Ramachandran V, Javeed N, Arumugam T, Dutta S, Klee GG, Klee EW, Smyrk TC, Bamlet W, Han JJ, Rumie Vittar NB, de Andrade M, Mukhopadhyay D, Petersen GM, Fernandez-Zapico ME, Logsdon CD, Chari ST. Adrenomedullin is up-regulated in patients with pancreatic cancer and causes insulin resistance in beta cells and mice. Gastroenterology. 2012 Dec;143(6):1510-1517.e1. doi: 10.1053/j.gastro.2012.08.044. Epub 2012 Sep 6. PMID 22960655
- [Derived] Antolino L, Rocca M, Todde F, Catarinozzi E, Aurello P, Bollanti L, Ramacciato G, D'Angelo F. Can pancreatic cancer be detected by adrenomedullin in patients with new-onset diabetes? The PaCANOD cohort study protocol. Tumori. 2018 Aug;104(4):312-314. doi: 10.5301/tj.5000693. Epub 2018 May 8. PMID 29192743